CLINICAL TRIAL: NCT06874777
Title: Effect of Aromatherapy Applied by Inhalation on Anxiety and Fatigue Levels in Individuals With Implantable Cardioverter Defibrillator (ICD)
Brief Title: Implantable Cardioverter Defibrillator (ICD) Patients and Inhalation Aromatherapy
Acronym: ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sebiha Aktaş Us, Nurse specialist/PhD student, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Erciyes
Record Dates: First submitted 2025-02-27; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Implantable Cardioverter Defibrillator (ICD); Aromatherapy; Anxiety; Fatigue Symptom
Keywords: Aromatherapy; anxiety; implantable cardioverter defibrillator (ICD); nursing; fatigue
MeSH Terms: conditions — Anxiety Disorders; Fatigue

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aromatherapy group (Experimental): Each participant in the intervention group was provided with lavender oil inhalation in addition to their routine treatments within the framework of the application protocol. This was administered by two surveyors, instructing the patients to apply it themselves. The method involved placing two drops of lavender oil on a gauze pad, holding it 5 cm below the nose for two minutes, followed by three deep breaths. This procedure was carried out for one month.
  Interventions: Other: Aromatherapy group
- control group (No Intervention): The control group was provided with routine treatment

INTERVENTIONS:
Other: Aromatherapy group — It is known that aromatherapy is used in symptom management in chronic diseases. When the literature is examined, it is seen that aromatherapy application is effective in relieving anxiety and fatigue in cardiovascular diseases. Currently, there is no symptom management method other than pharmacological treatment that is widely used or recommended by health professionals for ICD patients. The literature review reveals that there is no study examining the effect of lavender oil aromatherapy in relieving anxiety and fatigue in individuals with ICD implantation. In this context, the aim of this study is to determine the effect of aromatherapy applied by inhaling two drops for two minutes before going to bed for one month on anxiety and fatigue levels in individuals with ICD implantation.
  Other Names: Aromatherapy inhalation
  Arms: aromatherapy group

SUMMARY:
The effective management of anxiety and fatigue, which lead to negative physical, social, and psychological impacts and increase treatment costs in individuals with implanted cardioverter-defibrillators (ICD), is of great importance. Complementary and integrative therapy (CIT) methods offer a non-pharmacological, easy-to-apply, and safe intervention alternative for nurses and patients experiencing these symptoms. This study was conducted to investigate the effect of lavender oil aromatherapy, applied by inhalation for two minutes with two drops before bedtime for one month, on anxiety and fatigue levels in individuals with ICD, in a randomized controlled single-blind study design. A total of 86 patients with ICD implantation were included in the study, and 43 patients were randomly assigned to the intervention and control groups. The intervention group received lavender aromatherapy for two minutes with two drops of lavender oil inhaled before bedtime every night for one month, in addition to their routine treatment. The control group received only routine treatment. The study was conducted after obtaining the necessary ethical approval, institutional permission, and informed consent from the patients. The Patient Diagnosis Form, Piper Fatigue Scale (PFS), Spielberger State-Trait Anxiety Inventory Short Form (STAI-SF and STAI-TF), and Visual Analogue Scale (VAS) for Fatigue were used in data collection. The data were analyzed using the Statistical Package for Social Sciences (SPSS) 25.0 and G*Power program. A value of p<0.05 was considered statistically significant in comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were willing to participate in the study,
* aged between 18 and 65 years,
* with no physical or mental health issues that would hinder communication,
* had an ICD implanted at least 6 months ago,
* had a battery life of at least 3 months,
* had a fatigue level of 3 or higher on the Visual Analog Scale for Fatigue (VAS-F),
* had an EF of 40% or higher,
* and were visiting the cardiology outpatient clinic for ICD control

Exclusion Criteria:

* Individuals receiving anxiolytic or antidepressant treatment,
* those with respiratory system diseases (such as asthma, bronchitis, or chronic obstructive pulmonary disease), 19,231 characters left
* those with a known sensitivity to the essential oils used, and individuals with an olfactory impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Change severity of fatigue | Within 1 month and at the end of the 1st month
  2-point changes in the Visual Analoque Scale Fatigue Scale (VAS-F). VAS is known to be used for assessing the severity of fatigue symptoms. The scale consists of a 10 cm ruler, with one end labeled as 0 - "I do not feel fatigued" and the other end labeled as 10 - "I feel extremely fatigued." A score of 0-3 indicates "mild fatigue," 4-6 indicates "moderate fatigue," and 7-10 indicates "severe fatigue." In the study, interviewers explained to the patients that the 0-10 scale represents the severity of fatigue, and they were asked to mark the point corresponding to their fatigue level with a pen.
Change level of fatigue | Within 1 month and at the end of the 1st month
  1-point change in the average score of the Piper Fatigue Scale.The scale is a 5-point Likert-type scale. As the score obtained from the scale increases, the level of fatigue also increases.

OTHER OUTCOMES:
Change level of anxiety | Within 1 month and at the end of the 1st month
  2-point changes in the average score of the State anxiety inventory Short Form 2-point changes in the average score of the Trait anxiety inventory Short Form. The inventory consists of a total of 10 items. The first 5 items measure state anxiety, while the second 5 items assess trait anxiety. In the first 5 items, which evaluate how a person feels "at the moment," participants are expected to choose one of the following options: (1) "not at all," (2) "sometimes," (3) "very much," and (4) "completely." Similarly, in the second 5 items, which also assess how a person feels "at the moment," participants are expected to select one of the following responses: (1) "almost never," (2) "sometimes," (3) "most of the time," and (4) "almost always." Individuals who score 10 or above on the State Anxiety Inventory-Short Form (SAI-SF) and 14 or above on the Trait Anxiety Inventory-Short Form (TAI-SF) are considered clinically anxious.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkish Ministry of Health, Adana City Training and Research Hospital, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Those are private personal informations

REFERENCES:
- [Background] Forman J, Baumbusch J, Jackson H, Lindenberg J, Shook A, Bashir J. Exploring the patients' experiences of living with a subcutaneous implantable cardioverter defibrillator. Eur J Cardiovasc Nurs. 2018 Dec;17(8):698-706. doi: 10.1177/1474515118777419. Epub 2018 May 18. PMID 29775072
- [Background] AlMohammed HI, A Alanazi N, Maghrabi EF, A Alotaibi M. Role of Aromatherapy as a Natural Complementary and Alternative Therapy in Cardiovascular Disease: A Comprehensive Systematic Review. Evid Based Complement Alternat Med. 2022 May 20;2022:4543078. doi: 10.1155/2022/4543078. eCollection 2022. PMID 35646155
- [Background] Gong M, Dong H, Tang Y, Huang W, Lu F. Effects of aromatherapy on anxiety: A meta-analysis of randomized controlled trials. J Affect Disord. 2020 Sep 1;274:1028-1040. doi: 10.1016/j.jad.2020.05.118. Epub 2020 May 26. PMID 32663929
- [Background] Hassanzadeh, M., Farsi, Z., & Sajadi, S. A. (2021). Comparison of the effect of Sedamin and aromatherapy with Lavender on fatigue severity of patients with heart failure: A three arm randomized controlled trial. Journal of Herbal Medicine, 30, 100514. https://doi.org/10.1016/j.hermed.2021.100514
- [Background] Karadag E, Samancioglu S, Ozden D, Bakir E. Effects of aromatherapy on sleep quality and anxiety of patients. Nurs Crit Care. 2017 Mar;22(2):105-112. doi: 10.1111/nicc.12198. Epub 2015 Jul 27. PMID 26211735
- [Background] Liu L, Liu R, Zhang L, Tang Y, Fan C. The effect of aromatherapy on patients with acute coronary syndrome: A systematic review and meta-analysis. Complement Ther Clin Pract. 2024 Nov;57:101882. doi: 10.1016/j.ctcp.2024.101882. Epub 2024 Jul 6. PMID 38976965
- [Background] Lopes, L. de S., Bündchen, D., Modesto, F. C., Quintão, M., Chermont, S., Cavalcanti, A. C. D., & Mesquita, E. T. (2020). Aromatherapy in Patients with Cardiovascular Diseases: A Systematic Review. International Journal of Cardiovascular Sciences. https://doi.org/10.36660/ijcs.20190086